CLINICAL TRIAL: NCT01481155
Title: Prospective, Single-center, Investigator-blinded, Randomized, Half-side, Comparative Study of Photodynamic Therapy vs. CO2 Laser Therapy in Treatment of Actinic Keratoses
Brief Title: Comparative Study of Photodynamic Therapy vs. CO2 Laser Therapy in Treatment of Actinic Keratoses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Dr. Nina Scola, Dr. med. Nina Scola, consultant in Ruhr University of Bochum, Ruhr University of Bochum
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PDT vs. CO2
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Actinic Keratosis
Keywords: actinic keratosis; field cancerisation
MeSH Terms: conditions — Keratosis, Actinic | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Investigator

INTERVENTIONS:
Procedure: ablative CO2 laser therapy — CO2 laser therapy
Procedure: photodynamic therapy — Treatment with 5-ALA cream, application time at least 4 h, red light radiation with 76 J/cm²

SUMMARY:
The purpose of this study is to determine whether photodynamic therapy or CO2 laser therapy is superior in the treatment of actinic keratoses with respect to efficacy and side effects.

DETAILED DESCRIPTION:
Ablative laser therapy and photodynamic therapy are widely used and accepted therapeutic methods to treat multiple actinic keratoses, yet comparative studies are rare. The purpose of this study is to compare both treatments intraindividually with respect to treatment efficacy and side effects.

ELIGIBILITY:
Inclusion Criteria:

* men and women with clinical and histological diagnosed, symmetrical distributed actinic keratoses
* at least 2 actinic keratoses, on each of both treatment areas at least one
* Patients must be 18 years or older.

Exclusion Criteria:

* Age 17 years or younger
* lack of patient's informed consent for any of the two treatments
* contraindication for Co2 therapy or for photodynamic therapy
* skin infection in the treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Number of actinic keratoses 3 months after treatment | 3 months

SECONDARY OUTCOMES:
Histologic features | 1 month after therapy
Epidermal thickness in optical coherence tomography | 1 month after therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Venereology and Allergology, Ruhr University, Bochum, Germany